CLINICAL TRIAL: NCT01606111
Title: A Randomized, Double-blind, Placebo-controlled Trial to Investigate Safety and Efficacy of Cerebrolysin in Patients With Traumatic Brain Injury
Brief Title: The CAPTAIN Trial: Cerebrolysin Asian Pacific Trial in Acute Brain Injury and Neurorecovery
Acronym: CAPTAIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor patient recruitment
Sponsor: Ever Neuro Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVE-CN-0610
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — cerebrolysin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% NaCl, saline (Placebo Comparator)
  Interventions: Drug: 0.9% NaCl, saline
- Cerebrolysin (Experimental)
  Interventions: Drug: Cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — IV infusion, 50 ml/day, 10 days (treatment cycle will be repeated one and two months later if patient has a score of less than 7 in the extended Glasgow Outcome Scale on Day 30)
  Other Names: Cognicer, Renacenz
  Arms: Cerebrolysin
Drug: 0.9% NaCl, saline — IV infusion, 50 ml/day, 10 days (treatment cycle will be repeated one and two months later if patient has a score of less than 7 in the extended Glasgow Outcome Scale on Day 30)
  Other Names: Saline
  Arms: 0.9% NaCl, saline

SUMMARY:
The purpose of this trial is to investigate safety and efficacy of Cerebrolysin as add-on therapy to standard care in patients with acute traumatic brain injury (TBI). The study duration for each patient is 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TBI and a GCS 7-12
* Only isolated TBI
* CT
* Pre-Trauma Karnofsky-Index = 100
* Age 18-60 years
* Male and female patients
* Time to needle for study medication within 6 hours after injury
* Patient is not pregnant or lactating during the trial and is not of childbearing potential
* Patient was able to speak, read and write in a pre-defined study language before the accident.
* Reasonable expectation of completion of outcome measures at follow-up
* Written informed consent

Exclusion Criteria:

* Evidence of pre-existing major health problems
* Any neurological or non-neurological condition independent from TBI that might influence the functional outcome or other efficacy outcome measures
* Injury of writing hand influencing cognitive or other outcome measures
* Clear clinical signs of intoxication influencing the evaluation
* Major drug dependency including alcohol
* Chronic treatment with steroids, Ca2+-channel blockers or major anticoagulants
* Penetrating high-velocity missile head trauma
* Stab wound trauma into the brain
* Patients with spinal cord injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of mean score in MMSE, PSI, Stroop Color-Word Test, Early Reha BI, GOS-E | Day 10
  Global status is assessed by an ensemble of appropriate, single efficacy criteria to be tested by a multivariate, directional test approach
Composite endpoint of mean score in PSI, Stroop Color-Word Test, Color Trails Test, Digit Span, Early Reha BI, Finger Tapping Test, MMSE, Hospital Anxiety and Depression Scale, GOS-E | Day 30
Composite endpoint of mean score in PSI, Stroop Color-Word Test, Color Trails Test, Digit Span, Early Reha BI, Finger Tapping Test, MMSE, Hospital Anxiety and Depression Scale, GOS-E | Day 90

SECONDARY OUTCOMES:
Mortality | Day 10
Mortality | Day 30
Mortality | Day 90
Composite endpoint of mean score in PSI, Stroop Color-Word Test, Color Trails Test, Digit Span, Early Reha BI, Finger Tapping Test, MMSE, Hospital Anxiety and Depression Scale, GOS-E | Day 180
Mortality | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Wai S Poon, Prof., Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Result] Poon W, Matula C, Vos PE, Muresanu DF, von Steinbuchel N, von Wild K, Homberg V, Wang E, Lee TMC, Strilciuc S, Vester JC. Safety and efficacy of Cerebrolysin in acute brain injury and neurorecovery: CAPTAIN I-a randomized, placebo-controlled, double-blind, Asian-Pacific trial. Neurol Sci. 2020 Feb;41(2):281-293. doi: 10.1007/s10072-019-04053-5. Epub 2019 Sep 7. PMID 31494820